CLINICAL TRIAL: NCT05905835
Title: Treatment of Symptomatic Drug Refractory Paroxysmal Atrial Fibrillation With the Synaptic Compliant Cryoablation Balloon and System
Brief Title: Treatment of PAF With the Synaptic System
Acronym: Sensation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Synaptic Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-0001
Record Dates: First submitted 2023-05-26; First posted 2023-06-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cryoablation Balloon (Experimental): The Synaptic Cryo Balloon will be used to isolate all targeted pulmonary veins.
  Interventions: Device: Synaptic Cryoablation System

INTERVENTIONS:
Device: Synaptic Cryoablation System — The Synaptic Cryo Balloon must be used to isolate all targeted pulmonary veins. Entrance block will be confirmed in all targeted pulmonary veins (PVs) after a 20-minute waiting period or provocative testing with adenosine or isoproterenol. Any additional ablation in the LA beside PV isolation is not allowed in this protocol. Additional ablation of the cavo-tricuspid isthmus (CTI) with a conventional market-approved RF catheter is allowed only in case a typical atrial flutter is documented in prior patient history or occurs during the case (either spontaneously or inducible).

SUMMARY:
Enrolled subjects will be treated with the Synaptic Cryoablation System. Treatment will include cryoablation of the pulmonary veins to achieve PVI. All subjects will be followed for twelve (12) months after completion of the index ablation procedure.

DETAILED DESCRIPTION:
A multi-center, open-label, prospective, single-arm, pre-market clinical study. Enrolled subjects will be treated with the Synaptic Cryoablation System. Treatment will include cryoablation of the pulmonary veins to achieve PVI. All subjects will be followed for twelve (12) months after completion of the index ablation procedure. Data will be collected at enrollment, procedure, discharge, 1, 3, 6 and 12- months to assess the safety and effectiveness of the System. Testing for recurrence of atrial fibrillation will include a 12-lead ECG at 1, 3, 6 and 12-months post-ablation, weekly event recorder transmissions (TTM) after the 3-month follow-up visit through the 12-month follow up, and a 24-h continuous Holter ECG recording at 6 and 12-months post ablation. Symptom triggered rhythm monitoring will be used throughout the effectiveness post-ablation period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of symptomatic Paroxysmal Atrial Fibrillation (PAF), defined as atrial fibrillation that terminates spontaneously or with intervention (either through procedure or drug therapy) within seven (7) days of onset. Minimum documentation includes the following:

  1. A physician's note indicating recurrent atrial fibrillation (AF) which includes at least two (2) symptomatic AF episodes within six (6) months prior to enrollment; AND
  2. One electrocardiographically (from any form of rhythm monitoring, including consumer devices) documented AF episode within 12 months prior to enrollment.
* Refractory or intolerant to at least one (1) Class I or III anti-arrhythmic medication or contraindicated to any class I or III medication.
* Suitable candidate for catheter ablation.
* Adults aged 18 - 80 years.
* Willing and able to comply with all baseline and follow-up evaluations for the full length of the study.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Diagnosis of persistent AF, i.e., continuous AF lasting longer than seven (7) days from onset
* In the opinion of the Investigator, any known contraindication to an atrial ablation or anticoagulation. Including but not limited to the identification of any atrial thrombus or evidence of sepsis
* History of previous left atrial ablation or surgical treatment for AF/AFL/AT
* Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause
* Body Mass Index (BMI) ≥ 40
* Structural heart disease or implanted devices as described below:

  1. Left ventricular ejection fraction (LVEF) < 40% based on most recent transthoracic echocardiography (TTE) or transesophageal echocardiography (TEE) performed ≤ 180 days prior to enrollment
  2. Left atrial diameter > 5.5 cm or left atrial volume > 50 ml/m2 indexed based on most recent TTE or TEE performed ≤ 180 days prior to enrollment
  3. Implanted pacemaker, ICD, CRT device within 90 days prior to enrollment
  4. Previous cardiac surgery, ventriculotomy, or atriotomy (excluding atriotomy for CABG)
  5. Previous cardiac valvular surgical or percutaneous procedure, or prosthetic valve, including mitral valve clips
  6. Interatrial baffle, closure device, patch, or patent foramen ovale (PFO) occluder
  7. Presence of a left atrial appendage occlusion device
  8. Presence of any pulmonary vein stents
  9. Coronary artery bypass graft (CABG), PTCA, PCI, or coronary stent procedures within 90 days prior to enrollment
  10. Unstable angina or ongoing myocardial ischemia
  11. ST-Elevation Myocardial Infarction (STEMI) within 90 days prior to enrollment
  12. Moderate or Severe Mitral Insufficiency or Mitral Stenosis, severity based on the most recent TTE or TEE performed ≤ 180 days prior to enrollment
  13. Evidence of left atrial thrombus
* History of cryoglobulinemia
* Significant untreated restrictive or obstructive pulmonary disease or chronic respiratory condition
* Renal failure requiring dialysis
* History of blood clotting or bleeding disease
* History of documented cerebral infarct, TIA or systemic embolism,excluding post-operative deep vein thrombosis (DVT) ≤ 180 days prior to enrollment
* Active systemic infection
* Pregnant or lactating (current or anticipated during the study)
* Current enrollment in any other study protocol where testing or results from that study may interfere with the procedure or outcome measurements for this study
* Any other condition that, in the judgment of the Investigator, makes the patient a poor candidate for this procedure, the study or compliance with the protocol (includes, but not limited to, vulnerable patient population, mental illness, Gastroesophageal Reflux Disease (GERD), addictive disease, terminal illness with a life expectancy of less than two (2) years, or extensive travel away from the research center)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
safety - proportion of subjects who experienced device/procedure related Major Adverse Events (MAEs) | 6 months
  The primary endpoint for safety is an analysis of the proportion of subjects who experienced device/procedure related Major Adverse Events (MAEs) that occur during the procedure or through the 6-month follow-up of the study. MAEs include any of the major complications as defined in the 2017 HRS expert consensus statement
Effectiveness | 12 months
  The primary effectiveness endpoint is freedom from documented recurrence of AF, atrial tachycardia (AT), or atrial flutter (AFL) based on electrocardiographic data through 12-month follow-up and excluding a 90- day blanking period.

SECONDARY OUTCOMES:
Safety - Incidence of early onset (within 7 days of the index ablation procedure) of serious adverse events (SAEs) | 7 days
  Incidence of early onset (within 7 days of the index ablation procedure) of serious adverse events (SAEs)
Safety - Incidence of late onset (>7 days) of SAEs | 12 months
  Incidence of late onset (>7 days) of SAEs
Safety - Change from baseline NIH Stroke Scale post-ablation | Day 1
  Change from baseline NIH Stroke Scale post-ablation
Effectiveness - Rate of acute procedural success, defined as confirmation of entrance block in all targeted pulmonary veins | Day 0
  Rate of acute procedural success, defined as confirmation of entrance block in all targeted pulmonary veins
Effectiveness - Rate of pulmonary vein isolation on a per-vein basis | Day 0
  • Rate of pulmonary vein isolation on a per-vein basis
Effectiveness - Use of antiarrhythmic drugs (AADs) during the effectiveness evaluation period | 12 months
  Use of antiarrhythmic drugs (AADs) during the effectiveness evaluation period
Effectiveness - Freedom from documented symptomatic AF or new onset of AFL/AT through 12-month follow-up and excluding the 90- day blanking period | 12 months
  Freedom from documented symptomatic AF or new onset of AFL/AT through 12-month follow-up and excluding the 90- day blanking period
Effectiveness - Freedom from documented symptomatic AF or new onset of AFL/AT off antiarrhythmic drug therapy through 12-month follow-up and excluding the 90-day blanking period | 12 months
  Freedom from documented symptomatic AF or new onset of AFL/AT off antiarrhythmic drug therapy through 12-month follow-up and excluding the 90-day blanking period
Effectiveness - Failure-free rate as defined in primary effectiveness endpoint at 6 months post procedure | 6 months
  Failure-free rate as defined in primary effectiveness endpoint at 6 months post procedure
Performance - Single procedure success defined as freedom from primary effectiveness failure without a repeat procedure | 12 months
  Single procedure success defined as freedom from primary effectiveness failure without a repeat procedure
Performance - Procedure time, defined as the time elapsed from first venous access to last sheath removal | Day 0
  Procedure time, defined as the time elapsed from first venous access to last sheath removal
Performance - Duration of LA dwell time, defined as time from the Cryo Balloon Catheter exiting the sheath in the LA to time of final PVI | Day 0
  Duration of LA dwell time, defined as time from the Cryo Balloon Catheter exiting the sheath in the LA to time of final PVI
Performance - Total cryoablation time for index procedure | Day 0
  Total cryoablation time for index procedure
Performance - Total fluoroscopy time for index procedure | Day 0
  Total fluoroscopy time for index procedure
Performance - Treatment time, defined as the time from the start of the first ablation delivery to the end of the last ablation delivery | Day 0
  Treatment time, defined as the time from the start of the first ablation delivery to the end of the last ablation delivery
Performance -Changes in the quality-of-life measures (AFEQT) between baseline and 12-month follow-up | 12 months
  Changes in the quality-of-life measures (AFEQT) between baseline and 12-month follow-up

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Banner University Medical Center, Phoenix, Arizona
  - Dignity Health Arizona Research Enterprise, Phoenix, Arizona
  - St. Bernard's Heart & Vascular, Jonesboro, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mercy General Hospital, Sacramento, California
  - St. Luke's Mid America, Kansas City, Missouri
  - Northwell Health - Lenox Hill Hospital, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Christus Health Frances Hospital, Tyler, Texas
  - VCU Pauley Heart Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No